CLINICAL TRIAL: NCT06892769
Title: The Effect of Postoperative Telehealth Counseling on Postoperative Recovery and Self-care Power in Geriatric Patients Undergoing Day Surgery
Brief Title: Effect of Postoperative Telehealth Counseling on Recovery and Self-Care in Geriatric Day Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Talhaoglu, Assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Geriatric surgery
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Geriatric Patient Care Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine care (No Intervention): Patients will only be called weekly to complete the scales.
- telehealth counseling application (Experimental): to provide active counseling by calling weekly by phone on issues that the patient needs
  Interventions: Other: telehealth counseling

INTERVENTIONS:
Other: telehealth counseling — Patients in the intervention group will be called every week (for 4 weeks) and will be trained in line with the determined guide and scales will be filled.
  Arms: telehealth counseling application

SUMMARY:
This study was planned as a randomized controlled experimental study to evaluate the effect of postoperative telehealth counseling on patient outcomes in geriatric patients undergoing day surgery.

Hypotheses of the Study H11: In geriatric patients undergoing day surgery, the postoperative self-care power of the intervention group receiving postoperative telehealth counseling is higher than the control group not receiving counseling.

H12: In geriatric patients undergoing day surgery, the postoperative recovery status of the intervention group receiving postoperative telehealth counseling is higher than that of the control group not receiving counseling.

Inclusion Criteria;

* 65 years of age or older,
* Having undergone day surgery (appendectomy, hernia operations, biopsy procedures, cholecystectomy...)
* No communication problems (no vision and hearing problems),
* No mental problems,
* Being able to communicate by telephone (by the patient or relative),
* Volunteering to participate in the study,
* Having at most two chronic diseases (Diabetes and Hypertension).

Exclusion Criteria;

* Surgery in emergency conditions,
* developed complications during the case

DETAILED DESCRIPTION:
Data Collection Forms Patient Information Form: The form, prepared by the researchers with the support of the literature, includes a total of twelve questions questioning sociodemographic characteristics (age, gender, educational status, marital status, smoking, alcohol use, comorbidity, height, weight, body mass index and surgical experience) and disease-related characteristics (surgical procedure performed) Postoperative Recovery Index (PRAI): TThe index consists of 5 sub-dimensions and 25 items. The sub-dimensions are psychological symptoms, physical activities, general symptoms, bowel symptoms and craving symptoms. When determining the sub-dimension score, the scores of the related items are summed and their arithmetic averages are taken. For the total score, all items are summed and the arithmetic mean is taken. Higher scores on the index reflect more difficulty in postoperative recovery, while lower scores indicate that postoperative recovery is easier. In Cengiz and Aygin's study, the Cronbach's alpha value of the ASIQ was determined as 0.96 (Cengiz, 2018).

Self-Care Power Scale: It was developed by Kearney and Fleischer in 1979. The scale, which is used to determine the ability and power of people to take care of themselves, consists of 35 statements (items). The maximum score is 140. The higher the score obtained from the scale, the higher the self-care or self-care ability and power of the individual. The cronbach alpha value of the scale is 0.92 Data Collection The investigator evaluated the patients admitted to the clinic with the decision of surgery according to the research criteria. The surgery date and intensive care processes of the patients planned to be included were followed. Patients who were visited in the clinic before discharge were verbally informed about the study in face-to-face interviews of 10-15 minutes with the patient's relatives in the room, and informed consent forms were signed. It was reported that the data would be collected by the researcher through face-to-face interviews.

* Patient identification form will be filled out
* Contact information (telephone) of the patients will be taken and contact information (telephone) of the researcher will be given to the patients/relatives
* Patients/relatives will be informed that they can receive telephone counseling services from the researcher for the problems they experience in home care processes
* In line with the "Discharge Training Guide" prepared by the researcher in line with the literature, discharge training will be given to the patients and their relatives once in the patient's room by meeting face-to-face for an average of 15-20 minutes.
* In the 1st and 4th week after discharge, patients will be called by the researcher by phone and counseling services will be provided again.
* Postoperative Recovery Index and Self-Care Power Scale will be completed every week. The study will be terminated in the 4th week.

Control Group Practices

* Patients who meet the sample selection criteria will be informed about the study and their verbal and written consent will be obtained by reading the voluntary information form
* Patient identification form will be filled out
* Contact information (telephone) of the patients will be obtained.
* In line with the "Discharge Training Guide" prepared by the researcher in line with the literature, discharge training will be given to the patients and their relatives once in the patient's room by meeting face to face for an average of 15-20 minutes.
* At the 1st and 4th week after discharge, the patients will be called by the researcher by phone and the Postoperative Recovery Index and Self-Care Power Scale will be filled out. The study will be finalized in the 4th week.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older,
* Having undergone day surgery (appendectomy, hernia operations, biopsy procedures, cholecystectomy...)
* No communication problems (no vision and hearing problems),
* No mental problems,
* Being able to communicate by telephone (by the patient or relative),
* Volunteering to participate in the study,
* Having at most two chronic diseases (Diabetes and Hypertension).

Exclusion Criteria:

* Surgery under emergency conditions,
* developed complications during the case

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperatıve recovery process | postoperative 1st, 2nd, 3rd, 4th week
  Data collection tools
  Postoperative Recovery Index (PRAI): The index consists of 5 sub-dimensions and 25 items. The sub-dimensions are psychological symptoms, physical activities, general symptoms, bowel symptoms and craving symptoms. When determining the sub-dimension score, the scores of the related items are summed and their arithmetic averages are taken. For the total score, all items are summed and the arith.
  Maximum Possible Score:
  If the scoring system for each item is on a scale (for example, 1 to 5), the maximum score for each sub-dimension would be the sum of the highest possible score for each item within that sub-dimension. The total maximum score is the sum of the maximum scores for all 25 items.
  If each item can score between 1 and 5, the maximum score per item is 5. Maximum score for 25 items: 5 x 25 = 125 (total score)
  Minimum Possible Score:
  The minimum score for each item is 1, so the lowest possible score for each sub-dimension is 25 (1 for each of the 25 ite